CLINICAL TRIAL: NCT04172064
Title: Myocardial Perfusion and Contractile Reserve in End-stage Renal Disease: A Prospective Study Combining Myocardial Perfusion Scintigraphy and Dobutamine Stress Echocardiography
Brief Title: Myocardial Perfusion and Contractile Reserve in End-stage Renal Disease
Status: Completed | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-564-f-S
Record Dates: First submitted 2019-11-19; First posted 2019-11-21 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: End-Stage Renal Disease; Cardiovascular Diseases
MeSH Terms: conditions — Kidney Failure, Chronic; Cardiovascular Diseases | interventions — Myocardial Perfusion Imaging; Echocardiography, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 377patients evaluated by MPS and DSE
  Interventions: Diagnostic Test: Myocardial perfusion scintigraphy

INTERVENTIONS:
Diagnostic Test: Myocardial perfusion scintigraphy
  Other Names: Dobutamine stress echocardiography

SUMMARY:
The investigators prospectively recruited a total of 377 ESRD patients evaluated for kidney transplantation between January 2010 and July 2013 in our centre. Criteria for participation were a GFR below 20 ml/min/1.73m² or the need for haemodialysis and an age ≥18 years. 323 patients were on regular dialysis, the remaining 54 patients were being prepared for impending dialysis. Patients with known ischemic heart disease were excluded from the study. All patients underwent a systematic analysis of cardiovascular risk factors based on structured interviews with a physician, health records, blood lipid levels, and routine MPS at rest and under stress. In addition, 230 ESRD patients (61%) received standardized DSE. Patients with signs of ischemia in MPS and/or DSE were evaluated for coronary angiography on clinical grounds.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is a critical condition and bears a high risk of cardiovascular events. However, clinical algorithms to identify patients with coronary vasculopathies are still not defined and standardized. Non-invasive imaging by myocardial perfusion scintigraphy (MPS) or dobutamine stress echocardiography (DSE) might be used in such patients, however, it is unclear if these provide complementary or identical information and how this correlates to coronary angiography. A direct comparison of these imaging approaches, excellently validated in coronary artery disease, has not yet been described in well-defined and large groups of ESRD patients.

The investigators therefore initiated a large prospective trial with 377 highly-selected and well-characterized end-stage renal disease patients without known coronary artery disease comparing the performance of standardized MPS and DSE. For the first time we here describe a significantly large proportion of ESRD patients with contradictory findings in MPS and DSE and its correlation to invasive coronary angiography hinting to complementary rather than identical information between both modalities. This is an excellent basis of future studies comparing the prognostic value of MPS versus DSE versus a combined MPS/DSE approach.

ELIGIBILITY:
Inclusion Criteria:

* GFR below 20 ml/min/1.73m²

Exclusion Criteria:

* children
* pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 377 ESRD patients evaluated for kidney transplantation between January 2010 and July 2013 in our centre. Criteria for participation were a GFR below 20 ml/min/1.73m² or the need for haemodialysis and an age ≥18 years. 323 patients were on regular dialysis, the remaining 54 patients were being prepared for impending dialysis. Patients with known ischemic heart disease were excluded from the study.
Sampling Method: Probability Sample
Enrollment: 377 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Ischemia | january 2010 - june 2013
  Number of patients with reversible perfusion defects in myocardial perfusion scintigraphy or wall motion abnormalities in stress echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Michael Schäfers, Prof., Principal Investigator — Department of Nuclear Medicine, University Hospital Münster

IPD SHARING:
Plan to Share IPD: No